CLINICAL TRIAL: NCT02753777
Title: Prevalence and Clinical Severity of Autoimmune Blistering Diseases
Brief Title: Autoimmune Blistering Diseases Study
Acronym: AIBD
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Victoria Werth, Professor of Dermatology, University of Pennsylvania
Other Study IDs: 824790
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Pemphigus Vulgaris; Pemphigus Foliaceus; Bullous Pemphigoid
MeSH Terms: conditions — Pemphigus; Pemphigoid, Bullous | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood specimens will be collected during regularly scheduled clinic visits. The specimens will be processed and stored at the research labs belonging to the principal investigator at the University of Pennsylvania and the Philadelphia VA Medical Center. The specimens will not be publicly available and will be coded and stored in a locked facility equipped with a freezer.
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: Questionnaires

SUMMARY:
Pemphigus and bullous pemphigoid (BP) are severe autoimmune blistering diseases (AIBD) that pose a critical need for new therapeutic approaches. Clinical trials in pemphigus and BP will require the availability of validated disease severity measures that can be used to define primary outcomes.

DETAILED DESCRIPTION:
The disease severity instruments for pemphigus and BP, the Pemphigus Disease Area Index (PDAI) and the Bullous Pemphigoid Disease Area Index (BPDAI), respectively, have the potential to capture changes in all grades of disease activity, including mild disease, and therefore represent a substantial improvement over simple lesion counts or measurements of affected body surface area. However, full validation of the PDAI and BPDAI for use in clinical trials will require additional and more extensive measurements that will enable us to classify patients correctly by disease severity and be able to define the minimal change in score that is clinically significant.

This database study will compare the Pemphigus Disease Area and Severity Index (PDAI) and the Bullous Pemphigoid Disease Area Index (BPDAI) against other disease severity measures, including the Autoimmune Bullous Skin Disorder Intensity Score (ABSIS) and a physician's global assessment. Additionally, patients will be asked to rate their overall disease severity using a visual analogue scale, the patient's global assessment. Participants will also have the option to donate blood samples to our AIBD blood bank for immunologic and pathophysiologic studies.

The purpose of this database study will also be to evaluate quality of life (QoL) measures and correlate these QoL measures with disease severity in patients with pemphigus and BP. QoL is an important and independent component of disease impact on patients. This database study will use the following QoL measures: the SF-36, which is a nonspecific QoL measure; the Skindez-29 and the Dermatology Life Quality Index (DLQI), which are dermatology-specific instruments; the Autoimmune Bullous Disease Quality of Life (ABQOL) and Treatment of Autoimmune Bullous Disease Quality of Life (TABQOL) questionnaires, which are AIBD-specific tools. The results will be utilized in planning future clinical studies.

The AIBD study will be conducted only at Penn at this time. Data from the study will be entered into a password protected, web-based database that is used only at Penn.

ELIGIBILITY:
Inclusion Criteria:

* Gender/Age: Males or females above 18 years old
* Diagnosis: pemphigus vulgaris, pemphigus foliaceus, bullous pemphigoid
* Subjects able to give informed consent

Exclusion Criteria:

* Patients who are under age 18 years.
* Patients without pemphigus or pemphigoid diseases
* Penn employees
* Penn students
* Cognitively impaired persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients over the age of 18 who have been diagnosed with pemphigus vulgaris, pemphigus foliaceus or bullous pemphigoid.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-04; Primary Completion 2030-01-02 (Estimated); Study Completion 2030-01-02 (Estimated)

PRIMARY OUTCOMES:
Pemphigus Disease Area Index (PDAI) | one year
Bullous Pemphigoid Disease Area Index (BPDAI) | one year

SECONDARY OUTCOMES:
Autoimmune Bullous Disease Quality of Life (ABQOL) | one year
Treatment of Autoimmune Bullous Disease Quality of Life (TABQOL) | one year
Autoimmune Bullous Skin Disorder Intensity Score (ABSIS) | one year

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Hospital of the University of Pennsylvania, Department of Dermatology, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania, Department of Dermatology, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No